CLINICAL TRIAL: NCT00843843
Title: Sleep Length and Circadian Regulation in Humans
Acronym: HAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Helen Burgess, Associate Professor, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HL083971; HL083971
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Sleep Disorders
Keywords: Circadian Rhythms
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 9 hour sleep, then 3 hour nap and 6 hour sleep (Active Comparator)
  Interventions: Device: Bright light box
- 3 hour nap and 6 hour sleep, then 9 hour sleep (Active Comparator)
  Interventions: Device: Bright light box

INTERVENTIONS:
Device: Bright light box — Bright light of about 5000 lux, administered while sitting at a desk.

SUMMARY:
This research will examine why sleep restriction reduces the body clock's response to bright light. The results will enable the optimization of the bright light treatment of people who suffer from circadian rhythm sleep disorders, which include shift work sleep disorder, jet lag, delayed sleep phase syndrome and winter depression, thereby improving public health and safety, well-being, mood, mental function, and quality of life.

DETAILED DESCRIPTION:
Millions of Americans suffer from circadian rhythm sleep disorders, which include shift work sleep disorder, jet lag, delayed sleep phase syndrome and possibly winter depression. These conditions are typically characterized by persistent insomnia and/or excessive daytime sleepiness, impaired performance, and gastrointestinal distress. These negative symptoms result from a misalignment between the timing of the external social world and the timing of the internal circadian (body) clock. Circadian rhythm sleep disorders are effectively treated with bright light, which phase shifts the circadian clock, thereby realigning it with the timing of the external social world.

It is widely recognized that social influences have led to an increasing prevalence of sleep restriction in modern society. We recently demonstrated for the first time that short sleep episodes, when compared to long sleep episodes, markedly reduce phase advances to bright light. Thus when people cut their sleep short, they inadvertently reduce their circadian responsiveness to bright light. The mechanism(s) behind these reduced phase shifts to light are unknown. However, there are at least two aspects of short sleep episodes that could be responsible for this effect. First, short sleep episodes are associated with partial sleep deprivation. Second, as humans sleep with their eyes closed and are usually exposed to light when awake, short sleep episodes are also associated with short dark lengths. Our overall goal is to determine the biobehavioral mechanisms by which short sleep episodes impair phase shifts to bright light. Specific Aim 1 is to determine the effect of partial sleep deprivation on phase advances to light, while controlling for dark length. Specific Aim 2 is to determine the effect of short dark lengths on phase advances to light while minimizing sleep deprivation. We will estimate the timing of the human circadian clock by measuring salivary melatonin, a neuroendocrine hormone released from the pineal gland, and collecting measures of sleep via actigraphy, and sleepiness, mood, gastrointestinal distress and cognitive performance via computerized assessment.

Characterization of the separate effects of sleep deprivation and dark length on circadian phase shifts to light in humans is critical to understanding how humans respond to light during their daily life activities. Furthermore, the findings of this research will produce important and practical recommendations for avoiding decrements to phase shifts to light, thereby optimizing the bright light treatment of circadian rhythm sleep disorders, and thus improving public health and safety, well-being, mood, cognitive function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers

Exclusion Criteria:

* color blindness with the Ishihara test
* obese people (BMI > 30)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Burgess, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Biological Rhythms Research Laboratory, RUMC, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 9 Hour Sleep (3days), Then 3 Hour Nap and 6 Hour Sleep (3days): 9 hour sleep (3days), then 3 hour nap and 6 hour sleep (3days). Each 3 day intervention included a morning bright light treatment of about 5000 lux, administered while sitting at a desk.
- 3 Hour Nap and 6 Hour Sleep (3days), Then 9 Hour Sleep (3days): 3 hour nap and 6 hour sleep (3days), then 9 hour sleep (3days). Each 3 day intervention included a morning bright light treatment of about 5000 lux, administered while sitting at a desk.
Period: Overall Study
Arm/Group | 9 Hour Sleep (3days), Then 3 Hour Nap and 6 Hour Sleep (3days) | 3 Hour Nap and 6 Hour Sleep (3days), Then 9 Hour Sleep (3days)
Started | 8 | 8
Completed | 6 | 6
Not Completed | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- 3 Hour Nap and 6 Hour Sleep, Then 9 Hour Nap: Bright light box: Bright light of about 5000 lux, administered while sitting at a desk.
- Total: Total of all reporting groups
Arm/Group | 9 Hour Sleep, Then 3 Hour Nap and 6 Hour Sleep | 3 Hour Nap and 6 Hour Sleep, Then 9 Hour Nap | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (9.0) | 26.5 (5.8) | 28.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Dim Light Melatonin Onset (Hours)
Description: Gold standard marker of circadian timing
Time Frame: 12 days from baseline to final dim light melatonin onset
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 9 Hour Sleep | 3 Hour Nap and 6 Hour Sleep
Number analyzed (Participants) | 12 | 12
hours | 1.93 (0.98) | 0.80 (0.92)

2. Secondary Outcome: Psychomotor Vigilance
Description: Fastest 10% reaction time (msec)
Time Frame: after short or long nights
Population: Means
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | 9 Hour Sleep | 3 Hour Nap and 6 Hour Sleep
Number analyzed (Participants) | 12 | 12
msec | 215.15 (32.57) | 221.16 (33.56)

ADVERSE EVENTS:
Time Frame: Duration of study = 48 days
Description: Subjects were asked to contact research staff 24/7 if any adverse events occurred at home and were asked every day when in laboratory if any adverse events.
Groups:
- 9 Hour Sleep; 3 Hour Nap and 6 Hour Sleep: Bright light box: Bright light of about 5000 lux, administered while sitting at a desk.
Arm/Group | 9 Hour Sleep | 3 Hour Nap and 6 Hour Sleep
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No